CLINICAL TRIAL: NCT00891943
Title: A Randomised Controlled Trial of a One to One Weight Management Intervention in Primary Care
Brief Title: A Trial of One to One Weight Management in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: NHS Camden (Other Government)
Responsible Party: Ms Kiran Nanchahal, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: phpepw71; Sponsors number:PHPEPW71
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2009-04

CONDITIONS: Obesity; Overweight
Keywords: Obesity; Overweight; Randomised controlled trial; Primary Care; Weight; Cardiovascular Risk; Diabetes; Quality of life
MeSH Terms: conditions — Obesity; Overweight; Body Weight; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Structured lifestyle support (Other): Intervention group-structured lifestyle support.
  Interventions: Other: Structured lifestyle support
- Usual care for weight management (No Intervention): This is the control group, and they will receive "usual care" for weight management at their GP practice.

INTERVENTIONS:
Other: Structured lifestyle support — The intervention group will meet with a research nurse on 14 occasions over the 1 year research study, for structured lifestyle support, including dietary, physical activity and behavioral advice. They will also receive a pedometer.
  Arms: Structured lifestyle support

SUMMARY:
The purpose of this study is to conduct a randomised controlled trial to assess the sustained effects on weight, selected risk factors and sense of well-being of offering individualized weight management advice in the primary care setting to patients who wish to lose weight; and to identify the key factors influencing the success of the intervention.

DETAILED DESCRIPTION:
Primary care could make a substantial impact on the increasing prevalence of overweight and obesity and their associated adverse impact on health. The lack of a proven intervention may deter health professionals in primary care from providing support to their overweight patients as few obese people recall receiving weight control advice from a health professional.

In this study we aim to conduct a large scale randomised controlled trial to assess the effectiveness of a longer-term structured lifestyle support programme provided by a research nurse and the provision of pedometers compared to usual care in overweight/ obese adults who wish to lose weight. We will assess the degree of weight loss over a period of 12 months as well as related factors such as changes in waist circumference, quality of life and cost-effectiveness of the interventions.

The research is highly relevant to policy making at both national and local levels.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or over
* BMI ≥ 25 kg/m2
* GP confirmation

Exclusion Criteria:

* pregnant or lactating women
* patients with renal failure, pacemakers or cancer
* participating in other research affecting weight
* Ability to complete questionnaires
* Ability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Changes in weight, waist circumference and percent body fat at 12 months. | 12 months

SECONDARY OUTCOMES:
Weight, waist circumference, and percent body fat at 6 months. | 0 and 6 months
BMI, blood pressure, resting heart rate; obesity and weight related quality of life, Rosenberg measure of self-esteem changes at 12 months. | 0 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Nanchahal, MSc, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (2):
- United Kingdom (2):
  - London School of Hygiene and Tropical Medicine, London
  - Several GP practices in the Camden and Westminster area., London

REFERENCES:
- [Derived] Noble LM, Godfrey E, Al-Baba L, Baez G, Thorogood N, Nanchahal K. Treatment fidelity in the Camden Weight Loss (CAMWEL) intervention assessed from recordings of advisor-participant consultations. BMC Obes. 2018 Sep 10;5:24. doi: 10.1186/s40608-018-0203-7. eCollection 2018. PMID 30214815
- [Derived] McCambridge J, Sorhaindo A, Quirk A, Nanchahal K. Patient preferences and performance bias in a weight loss trial with a usual care arm. Patient Educ Couns. 2014 May;95(2):243-7. doi: 10.1016/j.pec.2014.01.003. Epub 2014 Jan 13. PMID 24492159
- [Derived] Nanchahal K, Power T, Holdsworth E, Hession M, Sorhaindo A, Griffiths U, Townsend J, Thorogood N, Haslam D, Kessel A, Ebrahim S, Kenward M, Haines A. A pragmatic randomised controlled trial in primary care of the Camden Weight Loss (CAMWEL) programme. BMJ Open. 2012 May 4;2(3):e000793. doi: 10.1136/bmjopen-2011-000793. Print 2012. PMID 22561352